CLINICAL TRIAL: NCT04241224
Title: A Prospective, Multicenter Atherectomy Study Showing Luminal Gain in Subjects With Peripheral Vascular Blockages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ra Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMS 103
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Peripheral Arterial Disease
Keywords: lower extremity Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Excimer Laser Photoablation (Experimental): Device: DABRA Laser System
  Patients with symptomatic peripheral vascular disease undergoing an endovascular revascularization procedure utilizing the DABRA Laser System.
  Interventions: Device: Atherectomy

INTERVENTIONS:
Device: Atherectomy — Endovascular treatment of peripheral arterial disease
  Other Names: DABRA Laser System

SUMMARY:
To evaluate the safety and effectiveness of the DABRA Laser System in the atherectomy of peripheral vascular stenoses.

ELIGIBILITY:
Participants must meet all of the inclusion criteria to participate in this study:

Inclusion Criteria

1. Ability and willingness to give written informed consent and comply with follow-up requirements
2. PAD with Rutherford Class 2-5
3. Stenotic lesion(s) in the peripheral vasculature
4. Subject is a candidate for atherectomy for infrainguinal peripheral artery disease

Angiographic Inclusion Criteria

1. Target vessel with documented stenosis by angiography ≥70% and ≤100% by angiography (as determined by Investigator)
2. Target vessel ≤ 3.0 mm in diameter
3. Target Lesion ≤ 25cm in length
4. The lesion to be treated is not severely calcified
5. Untreated ipsilateral iliac stenosis ≤70% (or tortuosity that might prevent advancing sheath to lesion) as applicable depending on access
6. No use of another atherectomy device in the same procedure
7. Treatment site is not located in a graft
8. Treatment site is not in, or distal to, a previously placed stent
9. No flow limiting dissection proximal, distal, or in the target lesion (prior to the use of the investigational device)

Participants meeting any of the exclusion criteria at the time of enrollment (index procedure/ intervention) will be excluded from study participation:

Exclusion Criteria

1. Age below 22 years
2. Pregnant, breastfeeding, planning to become pregnant. If women of reproductive capability will be enrolled, status will be assessed via pregnancy testing. Subject must agree to use effective birth control measures for duration of study. Pregnancy during study must be reported immediately.
3. Myocardial infarction (MI) ≤ 60 days prior to procedure
4. Cerebrovascular Accident (CVA) ≤ 60 days prior to procedure
5. Endovascular or surgical procedure ≤ 30 Days prior to procedure or a planned endovascular or surgical procedure within 30 days after the index procedure
6. Disorders or allergies precluding use of radiographic contrast including renal insufficiency severe enough to contraindicate use of radiographic contrast
7. Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated
8. Life expectancy ≤ 12 months
9. Patient is participating in another investigational drug or device study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Technical Success | At Index Procedure
  The Primary Efficacy Endpoint is the mean reduction in percent diameter stenosis in each subject's primary lesion following treatment with the DABRA Laser System and before any other treatment, as assessed by an independent Angiographic Core Laboratory.
Freedom from Major Adverse Events (MAE) | 30 Days
  Primary safety endpoint is freedom from Major Adverse Events, defined as all-cause mortality, unplanned major target limb amputation (at or above the ankle), clinically driven target limb revascularization (CD-TLR) at 30 Days, as classified by the Clinical Events Committee (CEC).

SECONDARY OUTCOMES:
Incidence of Target Lesion Revascularization (TLR) at 6 months | 6 months
  Clinically driven target lesion revascularization (TLR) at 6 months.
Reduction in Residual Diameter Stenosis | At Index Procedure
  Incidence of achieving a residual diameter percent stenosis of ≤ 50% in the primary lesion on the day of treatment, prior to any adjunctive therapy.
Rutherford Classification | 30 Days, 6 Months
  Change from baseline in Rutherford Category.
Change in Percent Diameter Stenosis | 30 Days, 6 Months
  Percent diameter stenosis and change from baseline in percent diameter stenosis as measured by Doppler Ultrasound and assessed by an independent core laboratory.
Vessel Patency | 30 Days, 6 Months
  Vessel patency as measured by Doppler ultrasound and assessed by an independent core laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Athar Ansari, MD, Study Chair
Locations (10):
- United States (10):
  - California Heart & Vascular Clinic, El Centro, California
  - Merced Vein & Vascular Center, Merced, California
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - Vascardio Heart and Vascular Institute, Hialeah, Florida
  - MIMIT Health, Chicago, Illinois
  - MIMIT Health, Glen Ellyn, Illinois
  - Eastlake Cardiovascular, Roseville, Michigan
  - South Texas Vascular Institute, Edinburg, Texas
  - Texas Tech University Health Sciences Center - Center for Cardiovascular Health, Lubbock, Texas
  - Laser Surgical Solutions, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No